CLINICAL TRIAL: NCT01633268
Title: Estimation of Brain Biomechanics Using MRI
Brief Title: Estimating Brain Biomechanics Using MRI
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 120139; 12-CC-0139
Record Dates: First submitted 2012-06-30; First posted 2012-07-04 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer; Traumatic Brain Injury; Brain Mapping; Craniocerebral Trauma; Magnetic Resonance Imaging
Keywords: MRI (Magnetic Resonance Imaging); Traumatic Brain Injury; Natural History
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy men and women aged 18-65

SUMMARY:
Objective: In this study we will develop and apply imaging techniques to perform the first three-dimensional (3-D) measurements of brain biomechanics during mild head movement in healthy human subjects. Biomechanics is the application of mechanics, or the physical principles in action when force is applied to an object, to the anatomical structure and/or function of organisms. Such techniques will be invaluable for building computational models of brain biomechanics, understanding variability of brain biomechanics across individual characteristics, such as age and sex, and determining brain sub-structures at risk for damage when movement of the head is accelerated, such as during a traumatic event.

Study Population: Measurements will be performed on 90 healthy men and women aged 18-65.

Design: We will build upon the model pioneered by our collaborator, Dr. Philip Bayly. The model places a human subject in a magnetic resonance (MR) scanner with one of two head support units that allows a specific range of motion. Each head support is latched such that it can be released by the subject, and results in either a rotation of the head of approximately 30 degrees or a flexion-extension of the head of approximately 4 degrees. Although both supports are weighted so that the motion is repeatable if the subject is relaxed, the subject can easily counteract the weight. The resulting acceleration/deceleration is small (in the range of normal activities, such as turning one's head during swimming) and has been validated and used in other human investigations of brain biomechanics. The subject repeats the motion multiple times during the MR scan under their own volition and desired pace to measure motion of the head and brain.

Outcome measures: This project is a pilot study evaluating the potential of extracting three-dimensional estimates of brain deformation, such as strain measurements, using MR imaging. A primary outcome of this project will be a fast MR acquisition sequence for measuring 3-D brain deformation. The sequence will be evaluated by applying the protocol to human subjects, followed by preliminary quantification of the reproducibility and stability of deformation measurements.

...

DETAILED DESCRIPTION:
Objective

In this study we will develop and apply imaging techniques to perform the first three-dimensional (3-D) measurements of brain biomechanics during mild head movement in healthy human subjects. Biomechanics is the application of mechanics, or the physical principles in action when force is applied to an object, to the anatomical structure and/or function of organisms. Such techniques will be invaluable for building computational models of brain biomechanics, understanding variability of brain biomechanics across individual characteristics, such as age and sex, and determining brain sub-structures at risk for damage when movement of the head is accelerated, such as during a traumatic event. Using the developed imaging techniques above, we will acquire a sufficient number of data sets to create templates of the average brain response and stiffness based on age and sex. Anonymized raw and processed data will be made publicly available to improve computational models of brain biomechanics.

Study Population

Measurements will be performed on 194 healthy men and women aged 18-65.

Design

We will build upon the model pioneered by our collaborator, Dr. Philip Bayly. The model places a human subject in a magnetic resonance (MR) scanner with one of two head support units that allows a specific range of motion. Each head support is latched such that it can be released by the subject, and results in either a rotation of the head of approximately 30 degrees or a flexion-extension of the head of approximately 4 degrees. Although both supports are weighted so that the motion is repeatable if the subject is relaxed, the subject can easily counteract the weight. The resulting acceleration/deceleration is small (in the range of normal activities, such as turning one's head during swimming) and has been validated and used in other human investigations of brain biomechanics. The subject repeats the motion multiple times during the MR scan under their own volition and desired pace to measure motion of the head and brain. Additionally, we will use a type of MRI called magnetic resonance elastography (MRE), which measures brain motion in response to mild head vibration, to investigate brain stiffness.

Outcome measures

This project is a study evaluating the potential of extracting three-dimensional estimates of brain deformation, such as strain measurements and stiffness, using MR imaging. A primary outcome of this project will be MRI techniques for characterizing 3-D brain biomechanics. The techniques will be evaluated by applying the protocol to human subjects, followed by preliminary quantification of the reproducibility and stability of deformation and stiffness measurements. Acquired data will be made publicly available for use by the research community.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Between 18 and 65 years of age
* Able to provide written informed consent
* Able to lie flat for up to 2 hours
* Able to move head up to 220 times within 45 minutes without discomfort
* Good general health based on History and Physical (H&P) or History and Assessment (H&A)

EXCLUSION CRITERIA:

* Contra-indications to MRI scanning without contrast based on RADIS department MRI safety questionnaire
* Pregnancy
* Inner ear problems causing vertigo
* History of spinal cord injury, head injury or other musculoskeletal condition that may result in an aversion to or difficulty with turning one s head multiple times in succession
* Claustrophobia (no sedation is permitted under this protocol)
* Weight more than 250 lbs
* Height greater than 6'4"
* All employees/staff supervised by the Principle Investigator or Lead Associate Investigator are excluded from participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers between age 18 and 65.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-07-04 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
technical development of a method for providing three-dimensional measurements of brain biomechanics in vivo using MR imaging. | Day 1 of study
  Primary outcome of this project will be a fast MR acquisition sequence for measuring 3-D brain deformation. The sequence will be evaluated by applying the protocol to human subjects, followed by preliminary quantification of the reproducibility and stability of deformation measurements

SECONDARY OUTCOMES:
Measure of preliminary database of brain deformation | End of study
  A preliminary database of brain deformation measurements from a healthy cohort will allow initial characterization of the variability of brain response across sex and age.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are working on deciding if we will share IPD.

REFERENCES:
- [Background] Allen ME, Weir-Jones I, Motiuk DR, Flewin KR, Goring RD, Kobetitch R, Broadhurst A. Acceleration perturbations of daily living. A comparison to 'whiplash'. Spine (Phila Pa 1976). 1994 Jun 1;19(11):1285-90. doi: 10.1097/00007632-199405310-00017. PMID 8073323
- [Background] Bayly PV, Cohen TS, Leister EP, Ajo D, Leuthardt EC, Genin GM. Deformation of the human brain induced by mild acceleration. J Neurotrauma. 2005 Aug;22(8):845-56. doi: 10.1089/neu.2005.22.845. PMID 16083352
- [Background] Brun CC, Lepore N, Pennec X, Lee AD, Barysheva M, Madsen SK, Avedissian C, Chou YY, de Zubicaray GI, McMahon KL, Wright MJ, Toga AW, Thompson PM. Mapping the regional influence of genetics on brain structure variability--a tensor-based morphometry study. Neuroimage. 2009 Oct 15;48(1):37-49. doi: 10.1016/j.neuroimage.2009.05.022. Epub 2009 May 14. PMID 19446645
- [Derived] Gomez AD, Bayly PV, Butman JA, Pham DL, Prince JL, Knutsen AK. Group characterization of impact-induced, in vivo human brain kinematics. J R Soc Interface. 2021 Jun;18(179):20210251. doi: 10.1098/rsif.2021.0251. Epub 2021 Jun 23. PMID 34157896
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-CC-0139.html